CLINICAL TRIAL: NCT01333293
Title: The Effect of Xolair ® (Omalizumab) in Mastocytosis Patients Prospective Double-blind, Placebo-controlled, Multicentre Study, XOLMA-Study
Brief Title: The Effect of Xolair ® (Omalizumab) in Mastocytosis Patients
Acronym: XOLMA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025ACH03T V1
Record Dates: First submitted 2009-07-20; First posted 2011-04-11 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Mastocytosis
Keywords: mastocytosis; omalizumab
MeSH Terms: conditions — Mastocytosis | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental)
  Interventions: Drug: injections
- Placebo (Placebo Comparator)
  Interventions: Drug: injections

INTERVENTIONS:
Drug: injections — subcutaneous injections

SUMMARY:
Patients with mastocytosis often suffer from associated symptoms such as nausea, vertigo, fatigue, urticaria, abdominal cramps, diarrhea or hypotension due to release of mediators by mast cells. These patients have also an increased frequency of anaphylactic/anaphylactoid reactions due to allergens such as hymenoptera or nonspecific stimuli such as contrast media, local anesthetics or analgesics. In addition, there is increased osteoporosis in mastocytosis patients due to the activity of mast cell mediators on osteoblasts and osteoclasts. Symptoms of mastocytosis respond poorly to treatment with antihistamines or other antiallergic drugs. There is currently no specific treatment for this disease with the exception of rare cases. There are, however, some case reports suggesting that omalizumab might decrease symptoms including hypotensive events.

The aim of the study is to investigate whether patients suffering from mastocytosis benefit from a 6 month course of omalizumab with regard to symptoms and quality of life and whether the applied in vitro and in vivo monitoring tools represent useful surrogate markers for the efficacy of omalizumab in patients with mastocytosis.

* Trial with medicinal product

DETAILED DESCRIPTION:
The study will take place as double-blind placebo controlled study. After a first a run-period of 2 months for all participants randomization (1:1) in two group will take place:

Group A: With omalizumab treatment for 6 months; dosage and administration schedule according to body weight and total IgE level (1/2 of the patients). Group B: Placebo (1/2 of the patients). After 4 months of treatment in both groups patients are encouraged to stop all drugs given to reduce mast cell related effects, mainly antihistaminics . In case that disturbing symptoms are reoccurring patients are allowed to restart these drugs. The evaluation will take place after 5 months of treatment.

Finally, a follow up visit 1 and 4 months after the study will take place.

ELIGIBILITY:
Inclusion criteria:

* Histological proven mastocytosis (cutaneous or systemic);
* Diagnosis made by one marrow unction and/or skin biopsy or other histological work up;
* Age: 18-70 years

Exclusion criteria

* Age <18 years;
* Known hypersensitivity to omalizumab or any of its components;
* History of cancer in previous 5 years;
* Patients with serious infections;
* Patients with active tuberculosis or undergoing anti-TB therapy;
* Patients currently treated with systemic immunosuppressive agents;
* Female patients who are pregnant or breast feeding;Contraception must be performed by a save reliable and accept method such as oral or implanted contraceptives, intravaginal or male preservatives or permanent methods such as tubal ligation.
* Patients with known positivity for human immunodeficiency virus (HIV). HIV screening will be performed by an HIV 1/2 Antibody-detection test.

Note: Specific immunotherapy for insect sting allergy is no exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reduction of mast-cell induced adverse events and symptoms as summarized and calculated from patient's main complaint score and AFIRM score. | 10 months

SECONDARY OUTCOMES:
Effect on the consumption or possibility to reduce mast-cell related drugs | 10 months
Effect on: - Lung function (FEV1), analysed by standard lung function measurements - blood pressure, - quantitative measurement of pressure-induced wheal and flare. | 10 months
Effect on in-vitro parameters (Tryptase levels, density of Fc-IgE-R expression on basophils, Platelet-Activation-Factor (PAF) and cysteinyl leukotriene LTC4) | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (3):
- Switzerland (3):
  - University Hospital Berne (Insel) and Zieglerspital Berne, Bern
  - Geneva University Hospitals and Medical Faculty of the University of Geneva, Geneva
  - Allergy Unit, Department of Dermatology, University Hospital Zurich, Zurich